CLINICAL TRIAL: NCT00131924
Title: Phase II Study of High-Dose Estrogen in Postmenopausal Women With Hormone Receptor-Positive Metastatic Breast Cancer After Failure of Sequential Endocrine Therapies
Brief Title: High-Dose Esterified Estrogens in Treating Postmenopausal Women With Metastatic Breast Cancer That Has Failed Previous Hormone Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data Monitoring Committee recommended closure due to poor accrual.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: NCI 03B5; NU-03B5
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Estrogens, Esterified (USP)

INTERVENTIONS:
Biological: esterified estrogens

SUMMARY:
RATIONALE: High doses of esterified estrogens may stop the growth of breast cancer cells that no longer respond to hormone therapy.

PURPOSE: This phase II trial is studying how well high-dose esterified estrogens work in treating postmenopausal women with metastatic breast cancer that has failed previous hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response rate in postmenopausal women with estrogen and/or progesterone receptor-positive metastatic breast cancer that has failed prior sequential endocrine therapy treated with high-dose esterified estrogens (Menest^®).

Secondary

* Determine time to disease progression in patients treated with this drug.
* Determine the toxic effects of this drug in these patients.

OUTLINE: Patients receive oral high-dose esterified estrogens (Menest^®) 3 times daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 2 months.

PROJECTED ACCRUAL: A total of 18-35 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic disease
* Documented disease progression

  * Must have received and subsequently failed (due to disease progression) ≥ 2 prior sequential endocrine therapies for treatment of metastatic breast cancer

    * Disease progression during adjuvant tamoxifen is considered 1 prior therapy
    * The 2 most recent treatments must have been endocrine agents
* At least 1 objective measurable disease parameter
* Brain metastases allowed provided both of the following criteria are met:

  * Brain metastases were previously treated AND are currently stable
  * Brain metastases are not the only site of metastatic disease
* Hormone receptor status

  * Estrogen and/or progesterone receptor-positive tumor

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Postmenopausal, as defined by any of the following:

  * At least 50 years of age with an intact uterus AND amenorrheic for the past 12 months
  * At least 50 years of age without a uterus AND follicle-stimulating hormone (FSH) level within postmenopausal range
  * Under 50 years of age and FSH level within postmenopausal range
  * Prior bilateral oophorectomy

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* Adequate hematologic function

Hepatic

* Adequate hepatic function
* Bilirubin ≤ 1.5 times upper limit of normal
* No history of hepatic adenoma

Renal

* Adequate renal function
* No history of hypercalcemia or severe hypocalcemia

Cardiovascular

* No history of thrombophlebitis or thromboembolic disorders associated with prior estrogen use
* No active thrombophlebitis or thromboembolic disorders
* No history of uncontrolled hypertension

Other

* Not pregnant
* No undiagnosed abnormal vaginal bleeding
* No other serious medical illness
* No psychiatric illness that would preclude giving informed consent
* No other invasive malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Prior chemotherapy for metastatic disease allowed
* Prior adjuvant chemotherapy allowed

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Prior radiotherapy allowed provided the only site of measurable disease was not irradiated

Surgery

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2004-03; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Clinical response rate

SECONDARY OUTCOMES:
Time to disease progression
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: William J. Gradishar, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States